CLINICAL TRIAL: NCT05500443
Title: The Effects of Menaquinone-7 Supplementation in Patients With Severe Coronary Calcifications
Brief Title: The DANish COronary DEcalcification (DANCODE) Trial
Acronym: DANCODE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Axel Diederichsen, Professor, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DANCODE
Record Dates: First submitted 2022-08-11; First posted 2022-08-15 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Coronary Artery Disease
Keywords: Vitamin K2; Double-blinded, randomized, placebo-controlled study; Coronary artery calcification; Coronary artery plaque; Cardiac events
MeSH Terms: conditions — Coronary Artery Disease; Cardiovascular Diseases | interventions — Vitamin K 2; menaquinone 7

STUDY DESIGN:
Intervention Model Description: Patients are randomly assigned in a 1:1 ratio to either daily oral supplementation with vitamin K2 (Menaquinone-7 (MK-7)) (720 μg/day, K2VITAL®Delta) and D (25 μg/day) or placebo for 24 months. Treatment of both groups will last for at least 24 months. To evaluate progression in CAC score, a non-contrast CT-scan is performed at baseline and after 12 and 24 months of follow-up.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The tablets have identical appearance, including taste, color, and size. The randomization-list is available to the data- and safety monitoring board, but patients, nurses, physicians and other data collectors are blinded to the allocation during the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active treatment (Experimental): Tablets with vitamin k2 (Menaquinone-7 (MK-7)) 720 μg/day
  Interventions: Dietary Supplement: Vitamin K2 (Menaquinone-7)
- Placebo (Placebo Comparator): Tablets with placebo
  Interventions: Dietary Supplement: Vitamin K2 (Menaquinone-7)

INTERVENTIONS:
Dietary Supplement: Vitamin K2 (Menaquinone-7) — Oral supplementation with vitamin K2 (Menaquinone-7 (MK-7)) 720 µg/day and D 25 µg/day

SUMMARY:
1. Abstract

Introduction Coronary artery calcification (CAC) and especially progression in CAC is a strong predictor of acute myocardial infarction and cardiovascular mortality. A substudy in the recent Danish study, AVADEC, suggested a protective role of supplementation with vitamin K2 and D in the development of CAC. This finding should be interpreted with caution, but the perspective is very interesting. In this study, we will examine the effect of the supplementation on progression of CAC in men and women with severe CAC. We hypothesize that the supplementation will slow down the calcification process.

Method and analysis In this multicenter and double-blinded placebo-controlled study, 400 men and women with CAC score ≥ 400 are randomized (1:1) to treatment with vitamin K2 (720 µg/day) and vitamin D (25 µg/day) or placebo treatment (no active treatment) for two years. Exclusion criteria are treatment with vitamin K antagonist or coagulation disorders. To evaluate CAC score, a non-contrast CT-scan is performed at baseline and repeated after 12 and 24 months of follow-up. Primary outcome is difference in CAC score from baseline to follow-up at two years. Intention-to-treat principle is used for all analyses.

Ethics and dissemination There are no reported adverse effects associated with the use of vitamin K2. Prior to inclusion, the protocol will be approved by the Regional Scientific Ethical Committee for Southern Denmark and the Data Protection Agency. It will be conducted in accordance with the Declaration of Helsinki. Positive as well as negative findings will be reported.

DETAILED DESCRIPTION:
2. Introduction Ischemic heart disease causes 19% and 20% of all deaths among men and women,respectively, thus prevention is of outmost importance. Ischaemic heart disease is often silent until symptoms of myocardial infarction. However, subclinical coronary artery disease is easily detected by non-contrast cardiac CT scans as coronary artery calcifications (CAC). CAC increases with age, and men have higher CAC scores than women. In a population, in which CAC is absent, there is a very low risk of future CVD, but as the CAC score increases, so does the risk of ischaemic heart disease. Thus, to prevent CVD, identification and treatment of individuals with severe CAC is important.

Vitamin K and the calcification process Vascular calciﬁcation is a slowly progressive process and caused by an imbalance between the mechanisms that promote and inhibit the deposition of calcium in the vessel wall, and vitamin K-dependent proteins play an essential role in this inhibition. The most familiar K vitamin is phylloquinone (vitamin K1), as it is essential in activation of several coagulation factors. Menaquinone (vitamin K2) is another very important vitamin K species. Vitamin K2 is deemed necessary for γ-carboxylation of proteins related to the inhibition of arterial calcification, i.e. matrix-Gla proteins (MGP). Without these activated proteins, the balance of cellular calcium uptake and the mineralization process in bone and blood vessels is impaired. The inhibiting process of the vitamin K-dependent proteins was originally showed by Luo et al. in 1997. In a mice model they described activated (carboxylated) MGP to be an important inhibitor of vascular calcification. Likewise, observational human studies suggest that long-term use of vitamin K antagonist (which inhibits carboxylation of MGP) is associated with both increased coronary- and extra-coronary vascular calciﬁcation. Furthermore, combined low vitamins K and D status has been associated with increased all-cause mortality risk compared with adequate vitamins K and D status.

No recommendations of vitamin K2 supplementation are available; however, as demonstrated in a randomized controlled trial there is a dose-dependent decrease of uncarboxylated MGP concentrations by vitamin K2 supplementation (180 µg/day, 360 µg/day or placebo). Thus, we know that the daily intake in the Western world is not sufficient to meet the request for a complete activation of MGP. Additionally, there is no documented toxicity for vitamin K1 or vitamin K2, and the WHO has set no upper tolerance level for vitamin K intake.

The effect of high-dose vitamin K2 supplementation (720 µg/day) and vitamin D (25 µg/day) on aortic valve progression was examined in the very recent AVADEC trial. Aortic valve calcification progression was non-significantly decreased, however seemed to slow down the progression of CAC in patients with severe CAC (score > 400). In addition, the number of cardiac events and all-cause death was significantly lower (unpublished results). As this was a secondary outcome, a confirmatory trial is requested.

2.1. Hypothesis In a randomized setup, we test the hypothesis that supplementation with vitamin K2 (720 µg/day) and vitamin D (25 µg/day) in comparison to placebo will reduce the progression of CAC in patients with severe CAC.

3. Methods 3.1. Trial design The study is a double-blinded, randomized, placebo-controlled study. 3.2. Participants Patients with a CAC score above 400 are eligible patients in DANCODE.

Exclusion criteria are:

• History of myocardial infarction or coronary revascularization

* History of venous thrombosis including pulmonary embolism
* Coagulation disorders
* Vitamin K antagonist use
* Disorders of calcium and phosphate metabolism (as primary hyperparathyroidism)
* Women of childbearing age (due to radiation issues)
* A life-expectancy < 5 years The study will take place at Danish hospitals, from 2023 to 2026. 3.3. Intervention Patients are randomly assigned in a 1:1 ratio to either daily oral supplementation with MK-7 (720 μg/day, K2VITAL®Delta) and D (25 μg/day) or placebo for 24 months. Treatment of both groups will last for at least 24 months. During this time, participants will visit our research unit five times, at 6-month intervals (Figure 1). To evaluate CAC score, we will perform a non-contrast CT-scan at baseline and after 12 and 24 months of follow-up.

Month 0 3 6 9 12 15 18 21 24 Informed consent X Medical interview X X X X X Web-based survey X X X X Biochemical measurements X X X X X Biobank X X X Non-contrast CT X X X Contrast CT X X Echocardiography X X Figure 1: Timeline and applied tests during the trial 3.4. Outcome The primary endpoint is the change in CAC score from baseline to 24-months follow-up.

Secondary endpoints are:

* Change in CAC score from baseline to 24 months in men and women, respectively
* Change in CAC score from baseline to 24 months in two pre-specified subgroups (baseline CAC score <1000 and ≥ 1000)
* Change in coronary plaque composition by contrast CT from baseline to 24 months
* Cardiac events (non-fatal myocardial infarction, coronary revascularization and cardiac death) during the follow-up period
* Change in calcifications in the aortic valve by non-contrast CT from baseline to 24 months
* Change in quality of life from baseline to 24 months.

Exploratory endpoint is:

* Change in MGP with different phosphorylation (p and dp) and carboxylation forms (c and uc).

Safety endpoints are:

• Death

* Cardiovascular events (myocardial infarction, coronary revascularization, heart valve surgery, stroke, significant aortic disease (dissection, rupture and surgery) and significant peripheral artery disease (thromboembolisms and surgery)
* Venous thromboembolism including pulmonary embolism
* Bleeding (including intracranial bleeding and hemorrhage associated with a drop in hemoglobin of ≥ 2mmol/l)
* Cancer, including solid and hematologic
* Significant deterioration in laboratory measurements (hemoglobin, creatinine (eGFR), natrium, potassium, calcium, magnesium, albumin, phosphate, alkaline phosphatase, parathyroid hormone or prothrombin time-international normalized ratio (PT-INR)).

3.5 Sample size We are planning a study of a continuous response variable from independent control and experimental subjects with 1 control per experimental subject. In the AVADEC trial, the mean (standard deviation) two year CAC progression among 182 men with CAC score ≥ 400 was 380 AU (330 AU) in the placebo group, and 288 AU (280 AU) in the intervention group. The joint standard deviation was 311 AU. If this is true in a population of men and women, inclusion of 180 experimental subjects and 180 control subjects are needed to be able to reject the null hypothesis that the population means of the experimental and control groups are equal with probability (power) 0.8. The Type I error probability associated with this test of this null hypothesis is 0.05 (two-sided). Accordingly, 360 subjects are needed. However, to comply with the uncertainty and to account for drop-out of 10%, 400 patients will be included. The sample size is based on two years of treatment.

3.6 Stratified randomization Randomization is performed by the pharmacy at Odense University Hospital. Based on a computer-generated assignment scheme the tablets will have a random number according to the sequential order.

3.7 Blinding The tablets have identical appearance, including taste, color, and size. The randomization-list is available to the data- and safety monitoring board, but patients, nurses, physicians and other data collectors are blinded to the allocation during the study.

3.8 Statistical methods We will use the intention-to-treat principle for all analyses. The primary endpoint (change in CAC score) will be presented as continuous variable. Additionally, the changes are analyzed in men and women, respectively, and in two pre-specified patient subgroups (CAC score 400-999 AU and ≥ 1000 AU, respectively). Primary hypothesis testing will be done hierarchically to maintain a closed testing procedure: only if the overall treatment effect is statistically significant, testing in CAC strata will be performed with confirmatory intent, otherwise solely for explorative reasons. Secondary endpoints include 1) change in coronary plaque composition by contrast CT; 2) cardiovascular events and mortality; 3) change in calcifications in the aortic valve by non-contrast CT; and 4) change in quality of life (see also Section 3.4).

We use general linear models (employing group, time point, and group x time point interaction) for the primary and for secondary endpoints as well as potential harms. Missing data will be treated as such; supplementary sensitivity analyses making use of imputed values under the missing at random assumption will be conducted for the primary analysis if more than 5% of expected data points are missing.

3.9. Patient and Public Involvement Patients and public were not involved in the design of study.

4. Organization The Steering Committee will consist of Professor Axel Diederichsen (PI, Department of Cardiology, OUH), PhD Kristian Øvrehus (Department of Cardiology, OUH), MD Selma Hasific (Department of Cardiology, OUH), Professor Lars Melholt Rasmussen (LMR, Department of Clinical Biochemistry and Pharmacology, OUH), and two from each screening site. All practical issues concerning the treatment and data sampling will be handled by the steering committee.

The data and safety monitoring board (DSMB) consists of the following experts: Professor in Cardiology Hans Mickley and Professor in Clinical Biostatistics in Diagnostic Research Oke Gerke. During the study, only the independent data and safety monitoring board will have access to the complete database including the randomization-list.

The data registration is performed via REDCap (Research Electronic Data Capture) with logging and secure storage directly on a server under Odense Patient data Explorative Network (OPEN), Region of Southern Denmark.

5. Publication Project results reporting the primary endpoint will be published in peer reviewed international journals. Positive as well as negative findings will be reported.

6. Feasibility Every year, approx. 13,000 patients with suspected angina pectoris are examined by cardiac-CT in the Western Denmark. All data, including baseline cardiovascular risk factors, history of ischemic heart disease and symptoms, scan characteristics, and results, including measurements of the CAC score, are collected prospectively in the Danish Heart Registry. Approx. 9% of the patients referred for Cardiac CT have CAC score ≥ 400 AU, and approx. 1/3 of these will undergo coronary revascularization within 3 months after the Cardiac CT. Thus, approx. 800 patients a year fulfill the inclusion criteria to participate in DANCODE. The DANCODE secretariat at OUH will identify the eligible patients in the Danish Heart Registry, and an invitation is send by mail to these patients. If a patient is interested, he/she is invited to the local site to discuss the trial with a study nurse. If he/she is willing to participate in the study, informed consent is obtained, and he/she is randomly assigned to the vitamin K2 or placebo group. Thus, we are able to identify enough participants.

7. Safety and Ethics We will use exactly the same tablets in DANCODE as we did in the AVADEC trial. Thus the active treatment is pure natural vitamin K2 720 µg and vitamin D 25 µg per day. This dose was well-tolerated with no difference in quality of life. Also, we observed no difference in number of participation who abandoned the study.

In accordance with the AVADEC trial, a Belgian dose-finding study using 360, 720 or 1080 µg of vitamin K2 thrice weekly for 8 weeks in chronic haemodialysis patients found no severe adverse effects. Vitamin K2 was well tolerated and did not cause a hypercoagulable state. Thus, there are no reported adverse effects associated with the use of vitamin K2.

Each patient will undergo three CT scans during the DANCODE study. Epidemiological studies do suggest that radiation exposure is associated with a slightly increased risk of cancer. No large studies involving medically exposed adult cohorts are available, but a linear no-threshold model has been considered. The average dose of one non-contrast cardiac CT scan is 1 mSv. Two additional contrast cardiac CT scans are performed (baseline and 24 months) with an average dose of 3 mSv each, thus at average the participants in DANCODE will receive 9 mSv (baseline: 4 mSv, 12 months: 1 mSv and 24 months: 4 mSv). For comparison, the annual background radiation dose in Denmark is 3 mSv, and the average annual limit for radiation workers is 20 mSv.

An independent DSMB will be established to perform ongoing safety surveillance. None of the DSMB-members are directly or indirectly involved in the coordination, execution or analysis of the study. The following is assessed: 1) severe adverse events (death, myocardial infarction, coronary revascularization, stroke, heart valve surgery and venous thromboembolism), and 2) laboratory measurements (creatinine (eGFR), natrium, potassium, calcium, magnesium, albumin, phosphate, alkaline phosphatase, parathyroid hormone and prothrombin time-international normalized ratio (PT-INR)). If there is a reason for concern, the DSMB can advise to interrupt the study for further analysis, and the study can be terminated prematurely if the number of severe adverse events is significantly higher in the treatment group versus the placebo group. This will be discussed in a meeting with the investigators and DSMB. The investigator will inform the subjects in case of interruption or termination of the study.

Subjects can leave the study at any time for any reason if they wish to do so, without any consequences. The investigator can decide to withdraw a subject from the study for urgent medical reasons or in case of demonstrable poor adherence to the study medication. This is assessed by interview and pill-count. If subjects are required to take vitamin K antagonist during the course of the study they will be withdrawn from DANCODE.

The protocol will be approved by the Regional Scientific Ethical Committee for Southern Denmark and the Data Protection Agency, and it will be conducted in accordance with the Declaration of Helsinki. According to the Danish Medicines Agency, vitamin K is a dietary supplement, and accordingly DANCODE is not a medical trial. Written informed consent is obtained from each participant. The study will be registered at clinicaltrials.gov.

8. Funding Private foundations and companies are sought for funding. We expect that study tablets, including placebo, are provided free of charge by Kappa Bioscience, Norway and Orkla Care, Denmark. The companies are not involved in the design, execution of the study, analysis of the data or reporting of results.

9. Discussion CAC and especially progression in CAC is a strong predictor of acute myocardial infarction and cardiovascular mortality. This study will examine the effect of vitamin K2 supplementation on progression of CAC in a randomized, placebo-controlled study. We hypothesize that vitamin K2 supplementation will slow down the progression of CAC. If positive effects are shown, a new treatment option may be available to prevent not only progression of CAC, but also ischemic heart disease. The result of this study are expected in 2026.

10. Applied tests during the study 10.1. Medical interview Baseline data will be obtained at first visit. At the subsequent visits, an interview is conducted and the following is evaluated: incident cardiovascular disease, chest pain, dyspnea and quality of life (EurQol 5D). A web-based survey is performed 3 months after each visit to support compliance and to evaluate possible side effects.

10.2. Laboratory Assessment Blood samples are obtained at every visit. Routine parameters include: hemoglobin, creatinine (eGFR), urea, sodium, potassium, calcium, magnesium, albumin, phosphate, alkaline phosphatase, parathyroid hormone and prothrombin time-international normalized ratio (PT-INR). Additionally, leukocytes, thrombocytes, lipid profile, hemoglobin A1c, alanine transaminase, lactate dehydrogenase, bilirubin, creatine kinase, troponin T and c-reactive protein are measured at first and last visit.

As a part of the study, 40 mL of blood from each of the participants will be collected at baseline, 12 and 24 month visit and centrifuged, labeled, and stored at -80°C in a biobank until serial testing. Vitamin D and dephosphorylated-undercarboxylated Matrix Gla-Protein (dp-ucMGP) are measured in the biobank samples after the last patient visit.

10.3. Multi-Slice Computed Tomography Scans Cardiac CT scans will be performed using a dedicated cardiac CT- scanner. A standard non-contrast as well as contrast scan is performed according to usual clinical care. To assess the CAC scores the following CT settings are used: 120 kV tube voltage, and a prospectively scan 300 ms after the QRS-complex. The scanning protocol during the contrast scan depends on the local CT scanner and the patient heart rate. In patients with a stable heart rate above 60 beats per minute, orally or intravenously β-blocker are administered until the heart rate is appropriate (if possible below 60), and a prospectively gated protocol is used. In patients with a heart rate > 70 bpm despite β-blocker pretreatment or in case of an irregular heart rhythm, a prospectively scan 200-400ms after the QRS-complex is performed. Additionally, sublingual nitrates are administered prior to the scan. 50-80 mL of contrast agent are injected into an antecubital vein at a rate of 6.0 mL/s followed by 60 mL intravenous saline (6.0 mL/s) using a dual-head power injector. Data acquisition parameters depends on the local CT scanner, but slice collimation will be below 0.6mm, gantry rotation time as fast as possible and a tube voltage of 70 or 120 kV depending on patients' weight.

All scans are send to and analyzed at the core lab, Odense University Hospital. CAC scores is measured by using the Agatston method by summing-up all spots of calcifications in the coronaries. The coronary artery tree will be analyzed for the presence and severity of CAD, according to the classiﬁcation of the American Heart Association 16-segment model. Coronary plaques are deﬁned as visible structures within or adjacent to the coronary artery lumen, which can be clearly distinguished from the vessel lumen and the surrounding pericardial tissue. All coronary segments ≥2 mm in diameter with plaque will be analyzed using a semi-automated software. Scans are analyzed by an experienced cardiologist.

11. Danish Appendix:

12. References http://www.ehnheart.org/images/CVD-statistics-report-August-2017.pdf (accessed 29 Marts 2022).

Gerke O, et al. Prevalence and extent of coronary artery calcification in the middle-aged and elderly population. Eur J Prev Cardiol. 2022 Feb 9;28(18):2048-2055.

Erbel R, et al. Coronary risk stratification, discrimination, and reclassification improvement based on quantification of subclinical coronary atherosclerosis: the Heinz Nixdorf Recall study. J Am Coll Cardiol 2010;56(17):1397-1406. doi: 10.1016/j.jacc.2010.06.030.

Polonsky TS, et al. Coronary artery calcium score and risk classification for coronary heart disease prediction. JAMA 2010;303(16):1610-1616. doi: 10.1001/jama.2010.461.

Rennenberg RJ, et al. Arterial calcifications. J Cell Mol Med 2010;14:2203-2210.

Danziger J, et al. Vitamin K-Dependent Protein Activity and Incident Ischemic Cardiovascular Disease: The Multi-Ethnic Study of Atherosclerosis. Arterioscler Thromb Vasc Biol 2016;36:1037-1042.

Viegas CS, et al. Gla-rich protein acts as a calcification inhibitor in the human cardiovascular system. Arterioscler Thromb Vasc Biol 2015;35:399-408.

Schurgers LJ, et al. Vitamin K-dependent carboxylation of matrix Gla-protein: a crucial switch to control ectopic mineralization. Trends Mol Med 2013;19:217-226.

Luo G, et al. Spontaneous calcification of arteries and cartilage in mice lacking matrix GLA protein. Nature 1997;386:78-81.

Rennenberg RJ, et al. Chronic coumarin treatment is associated with increased extracoronary arterial calcification in humans. Blood 2010;115:5121-5123.

Weijs B, et al. Patients using vitamin K antagonists show increased levels of coronary calcification: an observational study in low-risk atrial fibrillation patients. Eur Heart J 2011;32:2555-2562.

Schurgers LJ, et al. Vitamin K-antagonists accelerate atherosclerotic calcification and induce a vulnerable plaque phenotype. PLoS One 2012;7:e43229.

Chaikriangkrai K, et al. Prevalence and Implications of Subclinical Coronary Artery Disease in Patients With Atrial Fibrillation. Am J Cardiol 2015;116:1219-1223.

van Ballegooijen AJ et al. Combined low vitamin D and K status amplifies mortality risk: a prospective study. Eur J Nutr. 2021;60:1645-1654. doi: 10.1007/s00394-020-02352-8 Dalmeijer GW, et al. The effect of menaquinone-7 supplementation on circulating species of matrix Gla protein. Atherosclerosis 2012;225:397-402.

Pucaj K, et al. Safety and toxicological evaluation of a synthetic vitamin K2, menaquinone-7. Toxicol Mech Methods 2011;21:520-532.

Lindholt JS, et al. Effects of menaquinone-7 supplementation in patients with aortic valve calcification: study protocol for a randomised controlled trial.BMJ Open. 2018 Aug 23;8(8):e022019.

Diederichsen A et al. Vitamin K2 and D in patients with aortic valve calcification (AVADEC): a randomized double blinded clinical trial. Circulation. 2022. In press. Caluwe R, et al. Vitamin K2 supplementation in haemodialysis patients: a randomized dose-finding study. Nephrol Dial Transplant 2014;29:1385-1390.

Theuwissen E, Cranenburg EC, Knapen MH et al. Low-dose menaquinone-7 supplementation improved extra-hepatic vitamin K status, but had no effect on thrombin generation in healthy subjects. Br J Nutr 2012;108:1652-1657.

Pucaj K, Rasmussen H, Moller M, Preston T. Safety and toxicological evaluation of a synthetic vitamin K2, menaquinone-7. Toxicol Mech Methods 2011;21:520-532.

Preston DL, Ron E, Tokuoka S et al. Solid cancer incidence in atomic bomb survivors: 1958-1998. Radiat Res 2007;168:1-64.

Einstein AJ, Knuuti J. Cardiac imaging: does radiation matter? Eur Heart J 2012;33:573-578.

Budoff M, et al. Progression of coronary calcium and incident coronary heart disease events: MESA (Multi-Ethnic Study of Atherosclerosis). J Am Coll Cardiol. 2013 Mar 26;61(12):1231-9.

ELIGIBILITY:
Inclusion Criteria:

Coronary artery calcium (CAC) score above 400

Exclusion Criteria:

* History of myocardial infarction or coronary revascularization
* History of venous thrombosis including pulmonary embolism
* Coagulation disorders
* Vitamin K antagonist use
* Disorders of calcium and phosphate metabolism (as primary hyperparathyroidism)
* Women of childbearing age (due to radiation issues)
* A life-expectancy < 5 years

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2023-02-08 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
Coronary artery calcium (CAC) score, all participants | From baseline to 24-months follow-up
  Change in CAC score

SECONDARY OUTCOMES:
CAC score, men only | From baseline to 24-months follow-up
  Change in CAC score
CAC score, women only | From baseline to 24-months follow-up
  Change in CAC score
CAC score below 1000 at baseline, all | From baseline to 24-months follow-up
  Change in CAC score
CAC score above 1000 at baseline, all | From baseline to 24-months follow-up
  Change in CAC score
Coronary plaque burden | From baseline to 24-months follow-up
  Change in coronary plaque composition by contrast CT
Cardiac events | From baseline to 24-months follow-up
  Non-fatal myocardial infarction, coronary revascularization and cardiac death
Aortic valve calcification (AVC) score | From baseline to 24-months follow-up
  Change in AVC score

CONTACTS AND LOCATIONS:
Locations (3):
- Denmark (3):
  - Department of Cardiology, Odense University Hospital, Odense, Odense C
  - Department of Cardiology, Svendborg
  - Department of Cardiology, Vejle

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After primary endpoint is published
Access Criteria: Data are available on reasonable request

REFERENCES:
- [Derived] Hasific S, Ovrehus KA, Hosbond S, Lambrechtsen J, Kumarathurai P, Mejldal A, Ravn EJ, Rasmussen LM, Gerke O, Mickley H, Diederichsen A. Effects of vitamins K2 and D3 supplementation in patients with severe coronary artery calcification: a study protocol for a randomised controlled trial. BMJ Open. 2023 Jul 14;13(7):e073233. doi: 10.1136/bmjopen-2023-073233. PMID 37451735

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-02-24): https://cdn.clinicaltrials.gov/large-docs/43/NCT05500443/SAP_000.pdf